CLINICAL TRIAL: NCT01020201
Title: A Observational Cohort Study to Identify Risk Factors for Post Operative Nausea and Vomiting Following General Anesthesia in Female Patient Underwent Gynecological Operation
Brief Title: Risk Factors for Post Operative Nausea and Vomiting(PONV) in Patients Underwent Gynecological Operation Under General Anesthesia
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wei Mei, Associate Professor, Huazhong University of Science and Technology
Other Study IDs: TJHMZK01003
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Anesthesia, General; Elective Gynecological Operation; Chinese Female Patient; Adult
Keywords: Anesthesia, General; Elective Gynecological Operation; Chinese female patient; Adult

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PONV group: patients with postoperative nausea and vomiting
- Control group: patients without postoperative nausea and vomiting

SUMMARY:
Risk factors for postoperative nausea and vomiting(PONV) such as past history of PONV and/or motion sickness, non-smoking status, female gender, planned opiate use for post-operative analgesia were identified in white people. Whereas, risk factors for PONV in female patient with mongolian race were not clear. As a different life style and genetic background, new risk factors may associate with PONV in this population. The present study is a prospective cohort study to identify risk factors for PONV within 24 postoperative hours in chinese female patients underwent gynecology operative under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Chinese female patient

Exclusion Criteria:

* Unstable vital sign
* Patients under mechanical ventilation
* Patients under sedition (RASS=<-2)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients underwent gynecological operation under general anesthesia between 2009.02 and 2009.05.
Sampling Method: Non-Probability Sample
Enrollment: 774 (Actual)
Dates: Start 2009-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting | within 24 postoperative hours

SECONDARY OUTCOMES:
Incidence of postoperative shivering | within 24 postoperative hours
Postoperative pain score with Numerical Rating Scale (NRS-11) | within 24 postoperative hours
Time to full recovery of intestinal function | within 24 postoperative hours
Preoperative and postoperative fasting time | within 24 postoperative hours
Length of postoperative hospital stay and Length of hospital stay | before discharge
Total health care costs | before discharge
Postoperative delirium in recovery room | within PACU stay

CONTACTS AND LOCATIONS:
Overall Officials: Yuke Tian, M.D., PhD., Study Chair — Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology; Wei Mei, M.D., Study Director — Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China